CLINICAL TRIAL: NCT04383613
Title: Prone Positioning for Patients on General Medical Wards With COVID19: A Multicenter Pragmatic Randomized Trial [COVID-PRONE]
Brief Title: Prone Positioning for Patients on General Medical Wards With COVID19
Acronym: COVID-PRONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Sinai Health System (Other); Toronto General Hospital (Other); University Health Network, Toronto (Other); William Osler Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-1
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Covid-19; ARDS
MeSH Terms: conditions — COVID-19 | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, pragmatic, unblinded, 2-arm, parallel, randomized controlled trial.
Masking Description: The study will be unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRONE POSITIONING (Experimental): Patients in this arm will be instructed to lie on their stomach while they are in bed for 7 days or until the first of study hospital discharge or not requiring supplemental oxygen for >24 hours or study outcome.
  Interventions: Other: Prone positioning
- STANDARD OF CARE (No Intervention): Patients in this arm are not specifically instructed to lie on their stomach while they are in bed.

INTERVENTIONS:
Other: Prone positioning — The intervention is prone positioning (i.e., instructing a patient to lie on their stomach while they are in bed) for 7 days or until the first of study hospital discharge or not requiring supplemental oxygen for >24 hours or study outcome. Patients will be asked to aim for prone positioning four times per day for at least two hours each time, and will be encouraged to sleep on their stomach at night.
  Arms: PRONE POSITIONING

SUMMARY:
COVID-PRONE is a multicenter, pragmatic, unblinded, 2-arm, parallel, randomized controlled trial seeking to compare the pre-emptive prone positioning (i.e. encouraging patients to adopt a prone position before they require mechanical ventilation) to the control arm of standard care alone. Randomization will be stratified by site.

DETAILED DESCRIPTION:
COVID-PRONE is a multicenter, pragmatic, unblinded, 2-arm, parallel, randomized controlled trial. The intervention is not a medication or a medical device. Instead, the intervention is instructing patients to lie on their stomach while they are in bed.

Patients will be randomized to receive either standard-of-care or pre-emptive prone positioning while in bed plus standard of care. Randomization will be stratified by site. Patients randomized to prone positioning will be instructed to i) lie on their stomach supported by their arms and a pillow at the level of their shoulders and another pillow at the level of the pelvis, ii) immediately thereafter their oxygen saturation will be checked, iii) after a two hour period they can reposition to supine (but should be educated on the use of prone position and encouraged to adopt prone position as often as tolerated while in bed); the 2-hour period will be encouraged four times each day in addition to during sleep overnight.

Since there are limited data on the potential risks and benefits of prone positioning, a feasibility analysis will be performed after 30 patients are randomized to identify the rate of serious adverse events in the prone group (e.g., rate of pneumonia, death, intubation) and to understand the change in oxygenation as a result of prone positioning.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. COVID-19 infection is suspected by the treating clinician or confirmed by diagnostic test
3. Able to lie on their stomach with verbal instruction
4. Requiring supplemental oxygen less than or equal to 50% FiO2
5. Capable to make treatment related decisions
6. Hospitalized in the last 48 hours with suspected or confirmed COVID-19 infection or diagnosed for nosocomial infection in the last 48 hours during their hospital stay

Exclusion Criteria:

1. Inability to follow commands (e.g., delirium, dementia)
2. indication for mechanical ventilation (e.g., reduced level of consciousness, rapid clinical deterioration)
3. contraindication to prone positioning (spinal cord injury, unstable c-spine, pelvic fracture, unstable airway, open chest or abdomen, anterior chest tube, recent abdominal surgery in past 14 days)
4. patients on home CPAP (continue positive airway pressure)
5. transfer from ICU in past 72 hours
6. need for telemetry at the time of randomization
7. pregnant (i.e., more than 20 weeks)
8. body mass index above 40 kg/m2 (based on clinician's assessment)
9. Recently completed or plan for intrathoracic or intra-abdominal surgical procedure
10. severe hemoptysis
11. pace-maker inserted in past 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of in-hospital all-cause mortality, invasive or non-invasive mechanical ventilation, or need for FiO2 of 60% or more | From date of randomization until the date of in-hospital all-cause mortality, invasive or non-invasive mechanical ventilation, need for FiO2 of 60% or more, or date of hospital discharge, whichever came first, assessed up to 4 weeks

SECONDARY OUTCOMES:
Length of hospitalization | Up to 4 weeks [or until hospital discharge]
Adverse events of prone positioning (i.e., venous thromboembolism, pneumonia) | Up to 7 days [or until hospital discharge]
In-hospital all-cause mortality | From date of randomization until the date of in-hospital all-cause mortality or date of hospital discharge, whichever came first, assessed up to 4 weeks
Invasive or non-invasive mechanical ventilation | From date of randomization until the date of invasive or non-invasive mechanical ventilation, or date of hospital discharge, whichever came first, assessed up to 4 weeks
Need for FiO2 of 60% or more | From date of randomization until the date of need for FiO2 of 60% or more, or date of hospital discharge, whichever came first, assessed up to 4 weeks
Composite outcome of in-hospital all-cause mortality, invasive or non-invasive mechanical ventilation, or need for FiO2 of 60% or more assessed at 30 days, 90 days and 1 year | 30 days, 90 days and 1 year after randomization
Time spent in prone positioning among patients achieving the composite outcome of in-hospital all-cause mortality, invasive or non-invasive mechanical ventilation, or need for FiO2 of 60% or more | Up to 7 days

OTHER OUTCOMES:
Feasibility outcome: Change in oxygen saturation before and after prone positioning (to be measured for 72 hours beginning at the time of randomization), which will be calculated as: | 72 hours
  I) The ratio between the patient's oxygen saturation and the amount of oxygen they're inspiring, II) Sustained (i.e., more than 5 minutes) drop in oxygen saturation less than 88% in the prone position on the same oxygen therapy required to maintain a saturation of >92% in the supine position.
Feasibility outcome: Rate or serious adverse events | Up to 7 days
  Rate of serious adverse events as identified through routine care by the patient's attending physician (e.g., venous thromboembolism, pneumonia) or through objective testing (i.e., death, transfer to the intensive care unit). Notably, bacterial pneumonia will be pragmatically defined through the combination of a chest x-ray report identifying evidence of pneumonia and the receipt of antibiotics known to treat pneumonia
Feasibility outcome: Adherence to prone positioning | Day 3 and day 7
  The patients will be called on day 3 and 7. The research assistant/coordinator will ask the patient to estimate the number of hours spent in prone position.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fralick, MD, PhD, Principal Investigator — Sinai Health System; Fahad Razak, MD, MSc, Principal Investigator — St. Michael's Hospital (Unity Health Toronto); Amol Verma, MD, MPhil, Principal Investigator — St. Michael's Hospital (Unity Health Toronto)
Locations (8):
- Canada (8):
  - William Osler Health System, Brampton, Ontario
  - William Osler Health System, Etobicoke, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fralick M, Colacci M, Munshi L, Venus K, Fidler L, Hussein H, Britto K, Fowler R, da Costa BR, Dhalla I, Dunbar-Yaffe R, Branfield Day L, MacMillan TE, Zipursky J, Carpenter T, Tang T, Cooke A, Hensel R, Bregger M, Gordon A, Worndl E, Go S, Mandelzweig K, Castellucci LA, Tamming D, Razak F, Verma AA; COVID Prone Study Investigators. Prone positioning of patients with moderate hypoxaemia due to covid-19: multicentre pragmatic randomised trial (COVID-PRONE). BMJ. 2022 Mar 23;376:e068585. doi: 10.1136/bmj-2021-068585. PMID 35321918